CLINICAL TRIAL: NCT02424162
Title: Comparative Study of Two Multifocal Intraocular Lens With Different Add Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0837
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2.75 group (Experimental): Patients with 2.75 diopters multifocal intraocular lens
  Interventions: Device: +2.75 diopters multifocal intraocular lens
- 3.25 group (Active Comparator): Patients with +3.25 diopters multifocal intraocular lens
  Interventions: Device: +3.25 diopters multifocal intraocular lens

INTERVENTIONS:
Device: +2.75 diopters multifocal intraocular lens
  Arms: 2.75 group
Device: +3.25 diopters multifocal intraocular lens
  Arms: 3.25 group

SUMMARY:
This study will compare cataract patients with implantation of diffractive multifocal IOL with an additional power of +2.75 diopters (Group 1) and with +3.25 diopters (Group 2). Evaluations will be performed 1 and 3 months following cataract surgery, including measurement of uncorrected distance visual acuity (UDVA), refractive error (manifest refraction [MR]), and uncorrected near visual acuity (UNVA) at 33, 40, and 50 cm. At 3 months, internal aberrations and contrast sensitivity will be evaluated and subjects will complete a questionnaire on outcomes satisfaction, visual symptoms, and spectacle use.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18
* cataract patients with lens opacities classification higher than grade III
* patients who desire to be spectacle indepence for distance and near vision

Exclusion Criteria:

* previous ocular surgery or trauma
* presence of corneal opacities
* fundus abnormalities
* glaucoma
* uveitis
* amblyopia
* systemic disease
* posterior capsule rupture during cataract surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-11-11; Primary Completion 2015-11-03 (Actual); Study Completion 2015-11-03 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 3 months
  Uncorrected distance visual acuity and uncorrected near visual acuity

SECONDARY OUTCOMES:
Contrast sensitivity measured by the Functional Acuity Contrast Test (FACT) of the Optec 6500 view-in test system | 3 months
  Internal aberrations measured by the ray-tracing aberrometer and contrast sensitivity measured by the Functional Acuity Contrast Test (FACT) of the Optec 6500 view-in test system
internal aberration measured by the ray-tracing aberrometer | 3 months
  Internal aberrations measured by the ray-tracing aberrometer and contrast sensitivity measured by the Functional Acuity Contrast Test (FACT) of the Optec 6500 view-in test system

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea